CLINICAL TRIAL: NCT01550172
Title: Improving Dementia Caregiver Sleep & the Effect on Heart Disease Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Meredith Rowe, Meredeth A. Rowe, RN, PhD Professor and Lewis & Leona Hughes Endowed Chair, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6201111800; 1R01AG039495-01 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Caregivers of Persons With Dementia
Keywords: dementia caregivers; caregivers; Alzheimer's caregivers; caregiver sleep; heart disease risk; dementia; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep Behavioral Therapy A and NHMS (Experimental): Participants in this arm receive behavioral therapy A for insomnia and the night home monitoring system.
  Interventions: Behavioral: Sleep Behavioral Therapy A and NHMS
- Sleep Behavioral Therapy B and NHMS (Active Comparator): Participants in this arm receive sleep behavioral therapy B and the night home monitoring system.
  Interventions: Behavioral: Sleep Behavioral Therapy B and NHMS

INTERVENTIONS:
Behavioral: Sleep Behavioral Therapy A and NHMS — The night home monitoring system provides caregivers with reliable alerts and information regarding the whereabouts of the person with dementia during the night.
  Sleep behavioral therapy A uses a combination of cognitive exercises and behavior adjustments.
  Arms: Sleep Behavioral Therapy A and NHMS
Behavioral: Sleep Behavioral Therapy B and NHMS — The night home monitoring system (NHMS) provides caregivers with reliable alerts and information regarding the whereabouts of the person with dementia during the night.
  Sleep behavioral therapy B uses primarily behavioral adjustments.
  Arms: Sleep Behavioral Therapy B and NHMS

SUMMARY:
The purpose of the study is to determine whether a combined intervention of a night home monitoring system and cognitive-behavioral therapy for insomnia (CBTi) is effective in improving sleep in dementia caregivers who arise at night.

DETAILED DESCRIPTION:
Informal caregivers provide the majority of care for chronically ill adults, including persons with dementia. While these individuals provide a great benefit to the chronically ill relative, being a caregiver is associated with deleterious health consequences, including premature mortality and higher rates of coronary heart disease (CHD). Another common complaint among dementia caregivers is poor sleep, which has been connected to premature mortality and higher rates of CHD in noncaregiving adults. Currently no sleep therapies are empirically validated as effective for caregivers of persons with dementia (PWD), and since PWD often arise at night, improving caregiver sleep could be potentially hazardous as a sleeping caregiver cannot provide supervision during night awakenings. Our primary purpose is thus to determine whether a combined intervention is effective in improving sleep in caregivers of PWD who arise at night. The intervention consists of a night home monitoring system that provides reliable alerts to caregivers when PWD leave the bed and move through the house. While this system improved home safety for PWD, it did not affect caregiver sleep, so a more traditional sleep therapy will be added-cognitive-behavioral therapy for insomnia. In the proposed study, experimental participants will receive the night home monitoring system + CBTi; active comparator participants will receive the night home monitoring system and sleep behavioral therapy. Participants will remain in the study for 29 weeks, with 4 data collection points. We hypothesize experimental participants will have less time awake after going to bed, and improved sleep efficiency (percent time asleep while in bed). Sleep data will be collected for multiple nights using actigraphy and sleep diary. Our secondary research questions focus on the relationship between poor sleep and CHD. Both in adults and in dementia caregivers, there appears to be a link between poor sleep and abnormal levels on coronary heart disease biomarkers, and likely an increase in CHD with poor sleep. We aim to further explore this relationship as well as determine whether levels of biomarkers improve with improved sleep from the intervention. We propose to draw blood samples at 4 data collection points and measure a set of biomarkers indicative of CHD.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver for a relative who has been diagnosed by a physician with dementia or Alzheimer's disease.
* Persons with dementia sleep in the same location each night.
* Caregiver provides care for persons with dementia with nighttime activity that occurs at least one night/week.
* Caregiver meets the standard criteria for Insomnia.
* Caregiver sleep problems affect daytime functioning.
* If caregiver uses sleep medication, dose stable for 6 months.
* Caregiver Telephone Interview for Cognitive Status Score > 25.
* Caregiver does not require assistive devices to walk in the home at night.

Exclusion Criteria:

* Caregiver receives respite care at night the majority of the time.
* Caregiver has diagnosed sleep disorder.
* Caregiver uses CPAP at night
* Caregiver has chronic illness that requires frequent, weekly treatment/assessment by a healthcare provider.
* Current use of anticoagulant medication by the caregiver.
* Caregiver Sleep Apnea-Hypopnea Index (AHI) score > 10 or > 15 if pulse oximetry ≥ 88%.
* Caregiver shows evidence of Restless Leg Syndrome per the Cambridge-Hopkins Restless Leg Syndrome Questionnaire.
* Montreal Cognitive Assessment (MOCA) score < 26.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total Wake Time (TWT) | Week 27-28
  Actigraphy, using the Actiwatch2, will be used to measure objective sleep; We will collect data for 14-day periods using a 30-second epoch length to accurately capture night-to-night variability.
  Subjects will also complete a sleep diary for each day of actigraphic data collection, which will provide subjective sleep values of TWT. Data collected include bedtime, sleep start, number awakenings, minutes awake during night, wake time, out-of-bed time, minutes spent napping the previous day, and a sleep quality rating.
Sleep Efficiency (SE) | Week 27-28
  Actigraphy, using the Actiwatch2, will be used to measure objective sleep; We will collect data for 14-day periods using a 30-second epoch length to accurately capture night-to-night variability.
  Subjects will also complete a sleep diary for each day of actigraphic data collection, which will provide subjective sleep values of SE. Data collected include bedtime, sleep start, number awakenings, minutes awake during night, wake time, out-of-bed time, minutes spent napping the previous day, and a sleep quality rating.
Nighttime Injuries | Week 27-28
  The Caregiver will be asked about any PWD injuries that occurred since the last data collection point. Injuries will be coded according to the American National Standards method of recording injuries. The following data are collected: nature of injury; part of the body affected; object, substance, exposure, or bodily motion that caused the injury; event that directly resulted in the injury; and time and place of the injury's occurrence. An injury will be considered nighttime if the caregiver reported being asleep at the time the injury occurred.

SECONDARY OUTCOMES:
D-Dimer Levels | Week 27
  D-Dimer is a marker of coagulation activation and has been associated with coronary events. It has also been inversely associated with wake after sleep onset as well as poor sleep quality and low sleep efficiency. D-dimer is a byproduct of fibrinolysis which remains after a blood clot has been degraded. It consists of two cross linked fragments of fibrinogen. Elevated levels of D-dimer are a marker of thrombosis, as it might occur along atherosclerotic plaques in coronary blood vessels. D-dimer will be measured by monoclonal sandwich ELISA, which measures in the 3.9 - 250 ng/ml range.
Tissue Plasminogen Activator Levels | Week 27
  Tissue Plasminogen Activator is an endothelial lining protein that catalyzes the conversion of plasminogen into plasmin, which is responsible for the degradation of fibrin into soluble degradation products. Caregivers of PWD showed higher levels of TPA. A meta-analysis of cardiovascular disease risk and TPA indicated that levels greater than 13.5 ng/ml increased CVD risk by 50%.
C-reactive Protein (CRP) Levels | Week 27
  C-reactive protein (CRP) is a non-specific marker of inflammation shown in many studies to be elevated in AD caregivers and to be associated with poor sleep. High sensitivity CRP levels are consistently and independently associated with increased risk of cardiovascular events. HS-CRP will be measured by an ELISA.
Intercellular Adhesion Molecule-1 (ICAM-1) | Week 27
  Intercellular adhesion molecule-1 (ICAM-1) is found in leukocytes and endothelium and is involved in adhesion of leukocytes to and through the endothelium. ICAM-1 is stimulated by the proinflammatory cytokines. ICAM-1 may participate in atherogenesis by increasing monocyte transmigration into the arterial intima.
IL-6, and TNFα Levels | Week 27
  It is becoming apparent that sleep and immunity are strongly related and that impairments in sleep increase these circulating cytokine levels. Further, caregivers of Alzheimer's patients show both impaired sleep and elevated IL-6 and TNF-α. Levels of IL-6, IL-1, and TNF-α are partially controlled by sleep, and also regulate sleep and many aspects of the immune response. IL-6 and TNF-α are central mediators in the inflammatory process by regulating acute phase and coagulation protein, and inflammation plays a central role in the development and instability of atherosclerotic plaques.

CONTACTS AND LOCATIONS:
Overall Officials: Meredeth Rowe, RN, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Roth AJ, Curtis AF, Rowe MA, McCrae CS. Using Telehealth to Deliver Cognitive Behavioral Treatment of Insomnia to a Caregiver of a Person With Alzheimer's Disease. J Cogn Psychother. 2022 Feb 1;36(1):3-23. doi: 10.1891/JCPSY-D-20-00055. PMID 35121676